CLINICAL TRIAL: NCT02062320
Title: Establishment and Evaluation of a Post Caesarean Acute Pain Service
Brief Title: Establishment and Evaluation of a Post Caesarean Acute Pain Service (PCAPS)
Acronym: PCAPS
Status: Completed | Type: Observational
Sponsor: Brno University Hospital (Other)
Responsible Party: Principal Investigator, Petr Štourač, MD, MD, Ph.D., Brno University Hospital
Other Study IDs: NT13906-4/2012
Record Dates: First submitted 2014-02-11; First posted 2014-02-13 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: The Efficacy of Analgesic Methods After Caesarean Section
Keywords: Acute Pain Service; postoperative analgesia; Caesarean Section; non-opioid analgesia; opioid analgesia; epidural analgesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PRE-PCAPS: Parturients who underwent delivery by Caesarean Section in the period October 2009 - September 2010
- POST-PCAPS: Parturients who underwent delivery by Caesarean Section in the period November 2010 - October 2011.

SUMMARY:
The aim of this study is to compare the efficacy of analgesic methods after Caesarean Section before and after Post Caesarean Acute Pain Service establishing.

ELIGIBILITY:
Inclusion Criteria:

* Caesarean Section performed from October 2009 to October 2011 (study period)
* completed "Evaluation of postoperative analgesia after Caesarean Section" form.

Exclusion Criteria:

* Not completed "Standard Evaluation of postoperative analgesia after Caesarean Section" form.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We evaluated all patients undergoing delivery via Caesarean Section under anaesthesia in the period 10/2009 - 10/2011.
Sampling Method: Probability Sample
Enrollment: 407 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 72 hours after Caesarean Section (CS)
  Comparison of pain intensity (Visual Analogue Scale (VAS)) during the postoperative period (72 hours) between the two groups according to postoperative analgesic method and method of anaesthesia.

SECONDARY OUTCOMES:
VAS score above 4 | 72 hours after CS
  unsatisfactory pain relief
Additional Analgesic Requests (AAR) Count | 72 hours after CS
  Comparison of the average value of the AARs count in groups in the first 72 hours after CS
Analgesia related complication Rate | 72 hours after CS
  Analgesia related complications including hypotension, hypertension, tachycardia, bradycardia, hypoventilation were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Petr Štourač, MD, Ph.D., Study Director — Brno Faculty Hospital, departement of anesthesiology and intensive care medicine
Locations (1):
- Faculty Hospital Brno, Brno, South Moravian, Czechia

REFERENCES:
- [Background] Pan PH. Post cesarean delivery pain management: multimodal approach. Int J Obstet Anesth. 2006 Jul;15(3):185-8. doi: 10.1016/j.ijoa.2006.04.004. No abstract available. PMID 16798441
- [Background] Ismail S, Shahzad K, Shafiq F. Observational study to assess the effectiveness of postoperative pain management of patients undergoing elective cesarean section. J Anaesthesiol Clin Pharmacol. 2012 Jan;28(1):36-40. doi: 10.4103/0970-9185.92432. PMID 22345943
- [Background] Stourac P, Suchomelova H, Stodulkova M, Huser M, Krikava I, Janku P, Haklova O, Hakl L, Stoudek R, Gal R, Sevcik P. Comparison of parturient - controlled remifentanil with epidural bupivacain and sufentanil for labour analgesia: randomised controlled trial. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2014 Jun;158(2):227-32. doi: 10.5507/bp.2012.073. Epub 2012 Oct 31. PMID 23128818